CLINICAL TRIAL: NCT05379283
Title: Does Topical Lidocaine Decrease Sweat During Exercise in the Heat?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ENS2
Record Dates: First submitted 2022-05-11; First posted 2022-05-18 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Sweat Pore Closure
Keywords: thermoregulation, sweating, exercise
MeSH Terms: conditions — Motor Activity | interventions — Lidocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lidocaine pretreated skin (Experimental): one arm will be pretreated with lidocaine before exercise in the heat
  Interventions: Drug: Lidocaine; Other: control
- control skin (No Intervention): the other arm will act as the control condition

INTERVENTIONS:
Drug: Lidocaine — effect of lidocaine on sweat production during exercise in the heat
  Arms: lidocaine pretreated skin
Other: control — one arm will be pretreated with topical lidocaine, the other arm will not
  Arms: lidocaine pretreated skin

SUMMARY:
Subjects will walk on a treadmill at 3 mph and sweat will be collected from both forearms. One arm will be pretreated with topical lidocaine, and the other will act as the control.

DETAILED DESCRIPTION:
Subjects will walk on a treadmill at 3 mph and sweat will be collected from both forearms. One arm will be pretreated with topical lidocaine, and the other will act as the control. Sweat will be collected via macroducts attached to each arm. Sweat production on each arm will be compared using t-tests.

ELIGIBILITY:
Inclusion Criteria: 18-35 years of age -

Exclusion Criteria: pregnant females

-

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2022-05-15 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
volume of sweat produced during exercise following topical lidocaine | one hour of exercise
  Volume of sweat produced during exercise following tipocal lidocaine

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Buono, Principal Investigator — San Diego State University
Locations (1):
- San Diego State University, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No